CLINICAL TRIAL: NCT03510221
Title: Effects of Supplementation of Fruit Extract (Cranberry, Blueberry and Pomegranate) on Blood Pressure, Autonomic Balance, Insulin Resistance and Oxidative Stress in Hypertensive Patients
Brief Title: Effect of Antioxidant Supplementation on the Autonomic Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hyperox
Record Dates: First submitted 2018-03-29; First posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2016-01

CONDITIONS: Hypertension; Oxidative Stress; Autonomic Imbalance; Insulin Resistance
Keywords: Hypertension; Oxidative stress; Antioxidant; Autonomic imbalance; Insulin resistance; Cytokines
MeSH Terms: conditions — Hypertension; Insulin Resistance | interventions — Antioxidants

STUDY DESIGN:
Intervention Model Description: A group of hypertensive patients and a group of normotensive individuals
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antioxidants (Active Comparator): Subjects received 3 antioxidant capsules (1 capsule of blueberry + 1 capsule of cranberry + 1 capsule pomegranate - a day) during 4 weeks.
  Interventions: Dietary Supplement: Antioxidants capsules
- Placebo (Placebo Comparator): Subjects received 3 placebo capsules during 4 weeks.
  Interventions: Dietary Supplement: Antioxidants capsules

INTERVENTIONS:
Dietary Supplement: Antioxidants capsules — 1 capsule of cranberry, 1 capsule of blueberry, and 1 capsule of pomegranate extracts were offered during 4 weeks

SUMMARY:
Recent evidence suggests that there is a directly proportional relationship between diets with a high concentration of antioxidants and the reduction of blood pressure and the risk of cardiovascular events. However, there is a gap with regard to research on the effects of these diets on vascular function, especially in humans. The aim of this study was to evaluate the effect of antioxidant supplementation through the consumption of blueberry, cranberry and pomegranate extract capsules (1 of each per day), the effect of the autonomic balance in hypertensive and normotensive adults.

DETAILED DESCRIPTION:
A clinical trial was performed, with 60 individuals, 30 normotensive and 30 hypertensive patients. Participants were of both sex, aged between 18 and 60 years and Body Mass Index (BMI) less than 35 kg / m². Venous blood samples were collected after 12-hour fasting for biochemical measurements (glucose, total cholesterol and LDL-cholesterol, HDL-cholesterol, triglycerides, uric acid, sodium, potassium, urea, creatinine, insulin), and adiponectin , interleukin-4 (IL-4), interleukin-2β (IL-2β), monocyte chemoattractant protein-1 (MCP-1), leptin, C-reactive protein, tumor necrosis factor alpha (TNF-α), interleukin-6 and nitrotyrosine. An anthropometric evaluation was performed with measures of weight, height, waist circumference and cervical circumference. The hemodynamic evaluation was done through a non-invasive monitor. The study participants were divided into 2 different groups: Group A (normotensive) and Group B (hypertensive). The capsules for antioxidant supplementation were of blueberry, cranberry and pomegranate, being one capsule of each a day. Study participants received placebo capsules for 4 weeks and then received the fruit extract capsules (blueberry, cranberry and pomegranate), one capsule a day for 4 weeks. All tests were performed at baseline, after 4 and 8 weeks of intervention. The comparison between groups was performed with the Multiple Comparison Test (ANOVA). The research project was approved by the Ethics Committee for Analysis of Research Projects (CAPPesq) of the Hospital das Clinicas of the Faculty of Medicine of the University of Sao Paulo. Participation in the research was voluntary and all participants read and signed the consent form. The risk for the present participant was minimal.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of hypertension - group Hypertensives
* Healthy people - group Normotensive

Exclusion Criteria:

* Patients with glycated hemoglobin > 7%,
* Patients with a diagnosis of cardiovascular disease,
* Patients with LDL-cholesterol> 160 mg/dL (non-diabetics)
* Pregnant women,
* Cigarret smokers,
* Diabetics using more than one drug in addition to metformin,
* Patients with LDL-cholesterol> 130 mg/dL (non-diabetic using statin),
* LDL cholesterol ≥ 100 mg / dL (patients on statin),
* Patients with valvular heart disease,
* Pulmonary hypertension,
* Patients with collagen disease,
* Patients with type of cancer,
* Complex arrhythmia,
* Those patients with any chronic crippling pathology.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Effect of antioxidants on heart rate variability in 29 normotensive subjects and 30 hypertensive patients | 4 weeks
  Antioxidant supplementation should improve heart rate variability as a consequence of improved antioxidant capacity

SECONDARY OUTCOMES:
Effect of antioxidants on insulin resistance in 29 normotensive subjects and 30 hypertensive patients | 4 weeks
  Supplementation with antioxidants should improve insulin resistance
Effect of antioxidants on blood pressure in 29 normotensive subjects and 30 hypertensive patients | 4 weeks
  Supplementation with antioxidants should improve blood pressure
Effect of antioxidants on antioxidant capacity in 29 normotensive subjects and 30 hypertensive patients | 4 weeks
  Supplementation with antioxidants should improve antioxidant capacity